CLINICAL TRIAL: NCT05607914
Title: Comparison of Acute Effects of Percussion Massage Therapy and Static Stretching on Hamstring Flexibility
Brief Title: Effect of Percussion Massage on Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Pinar Yasar, research assisstant, Suleyman Demirel University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 72867572-050.01.04-31
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Massage; Hamstring Flexibility; Manual Therapies
Keywords: massage; static stretching; hamstring muscles; flexibilty
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- percussion massage group (Active Comparator): Applying the hypervolt device to the hamstring muscle with the hard ball head for 5 minutes
  Interventions: Procedure: percussion massage
- static stretching group (Active Comparator): Static stretching of the hamstring muscle for 5 minutes
  Interventions: Procedure: static stretching
- control group (No Intervention): no intervention

INTERVENTIONS:
Procedure: percussion massage — percussion massage to the dominant leg hamstring muscle for 5 minutes
  Other Names: vibration massage
  Arms: percussion massage group
Procedure: static stretching — Static stretching to the dominant hamstring muscle for 5 minutes
  Arms: static stretching group

SUMMARY:
Background and aim: Percussion massage, which is one of the applications to increase muscle flexibility, is a method that combines vibration and massage therapy elements. With its popularity in recent years, it is offered as an alternative to traditional methods that increase flexibility. The aim of this study is to examine the acute effect of percussion massage and static stretching exercise on hamstring flexibility.

Method: Individuals with active knee extension angle limited to at least 15 degree were included in the study, which was designed as a cross-over. Active Knee Extension test and Sit and Reach Test were performed before and after the interventions for the evaluation of hamstring flexibility. Participants were divided into 3 groups as percussion massage, static stretching and control groups, interventions were made with 3 days intervals and control measurements were taken.

DETAILED DESCRIPTION:
Active knee extansion test: In this test, which is used to evaluate hamstring flexibility in the sitting position, the participant was asked to sit on the edge of the bed and the hip-knee flexion angle was adjusted to 90 degree. For the measurement of active knee extension degree, a double-arm universal goniometer (Baseline Stainless Steel Goniometer; Fabrication Enterprises Inc., Elmsford, NY, USA) was placed on the lateral condyle of the femur and the participant was told to actively extend the knee to full extension. The angle at the end point of the movement was recorded.

sit and reach test: While sitting in a long sitting position with their knees straight and their bodies upright, the participants were asked to touch the soles of their bare feet to the assessment table. In this position, they were told to reach as far as they could reach on the coffee table with their elbows straight and palms facing the floor. By measuring the distance between the fingertip and the coffee table, those who could reach the table received "0" values, those who could reach beyond the table (+) cm and those who could not reach (-) cm. The best value after two measurements was recorded.

Static stretching procedure: For the static stretching exercise, the participant was asked to lie down in the supine position. The investigator had the dominant side passively flexed the hip to 90 degree, extending the knee to the end that could be tolerated. At the last point, it was waited for 30 seconds and then the hamstring muscle was relaxed and rested for 30 seconds. A total of 5 minutes of application was completed by doing 5 repetitions with 30 seconds of static stretching and 30 seconds of rest in each period.

percussion massage procedure: Hypervolt (Hyperice, California, US) device was applied to the dominant hamstring muscle for 5 minutes at 53 Hz frequency with the "hard ball" head. Semitendinosus and semimembranosus muscles were focused in the first 2.5 minutes of the massage treatment, and the biceps femoris muscle in the second 2.5 minutes. By paying attention to the equal amount of pressure applied throughout the massage, the massage was started from the medial side of the muscle in the first part of the application and the massage was completed by moving the device from distal to proximal and from proximal to distal in a straight line within 20 seconds. While passing to the last 2.5 minutes, the massage device was shifted laterally at the distal end of the muscle, and the application was made from distal to proximal and then distally. Thus, the massage for each muscle was started from the medial and ended laterally.

ELIGIBILITY:
Inclusion Criteria:

-Active knee extension limited to at least 15 degrees

Exclusion Criteria:

* Having a hamstring injury in the past two years
* Having neurological problems in the lower extremity and lumbar region
* participate in a similar study within the past year

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
knee range of motion measurement | 2 minutes
  measurement of maximum knee extension angle in sitting position
hamstring flexibility measurement | 2 minutes
  Evaluation of the flexibility of the hamstring muscle in the long sitting position

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Yasar, MsC, Principal Investigator — Suleyman Demirel University
Locations (1):
- Faculty of Health Sciences, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No